CLINICAL TRIAL: NCT07089303
Title: Ultra-high Field Multimodal and Multinuclear Neuroimaging Cohort Study of Alzheimer's Disease
Brief Title: Alzheimer's Disease Multinuclear Imaging Neuro-Enhanced Resolution (AD-MINER)
Acronym: AD-MINER
Status: Recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xin Lou, Director and Clinical Professor, Chinese PLA General Hospital
Other Study IDs: ADMINER-PLAGH-2025
Record Dates: First submitted 2025-07-20; First posted 2025-07-28 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment Due to Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CN
- MCI
- AD

SUMMARY:
This single-center prospective cohort study will enroll 750 participants (250 cognitively Normal (CN) individuals, 250 with mild cognitive impairment (MCI), and 250 with Alzheimer's disease (AD)). At baseline and at annual follow-ups, participants will undergo 3 Tesla (3 T) and 7 Tesla (7 T) multimodal magnetic resonance imaging (MRI) scans, blood biomarker testing, genotyping, and cognitive assessments to identify early imaging biomarkers and construct models of disease progression.

DETAILED DESCRIPTION:
This prospective, single-center cohort will enroll 750 participants (normal controls, MCI, and AD) for at least four years of follow-up. Using ultra-high field 7T multimodal and multinuclear (hydrogen-1 [¹H], sodium-23 [²³Na]) MRI, combined with plasma biomarkers and genetic data, the study aims to identify early neuroimaging biomarkers and clarify the clinical significance of sodium metabolic abnormalities in AD. Structural, functional, and sodium imaging data will be integrated with neuropsychological and blood-based markers, using artificial intelligence for early diagnosis and risk prediction. The study will address technical gaps in early detection and provide the first standardized 7T AD neuroimaging database for the Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Age 55-90 years (inclusive).
* Willing and able to participate in baseline assessment and longitudinal follow-up; voluntary provision of biospecimens and personal information, and commitment to complete all follow-up visits.
* Able to undergo MRI scanning (no contraindications to MRI).
* Group-specific cognitive criteria:

CN: No subjective memory complaints beyond age expectation (confirmed by study partner); MMSE score 26-30 (inclusive; exceptions permitted for participants with <8 years of education with principal investigator approval; CDR = 0, memory box = 0; Normal cognitive and daily functioning, no significant impairment.

MCI: Subject, partner, or physician reports subjective memory concerns; MMSE criteria same as CN group; CDR = 0.5 (memory box ≥0.5); General cognition and function relatively preserved; does not meet criteria for AD.

AD: Subject, partner, or physician reports subjective memory concerns; MMSE score <26 (inclusive; exceptions as above); CDR = 0.5 or 1.0; Meets National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) probable AD diagnostic criteria or 2024 National Institute on Aging-Alzheimer's Association (NIA-AA) criteria (e.g., positive Pittsburgh compound B (PIB) and tau).

Exclusion Criteria:

* Self-reported or MRI-detected major neurological diseases other than AD: including but not limited to stroke (cerebral hemorrhage, infarction), congenital intellectual disability, intracranial tumors, epilepsy, Parkinson's disease, Huntington's disease, normal pressure hydrocephalus, progressive supranuclear palsy, multiple sclerosis, severe head trauma with persistent deficits, etc.
* Severe psychiatric disorders (e.g., schizophrenia requiring medication control) or other known brain structural abnormalities.
* Significant organ failure (heart, liver, kidney, etc.), malignant tumors, or short life expectancy making completion of follow-up unlikely.
* Contraindications to MRI (e.g., claustrophobia, incompatible pacemaker, aneurysm clip, artificial heart valve, cochlear implant, or other metallic implants).
* Other clinical history or examination findings judged by investigators as potentially unsafe for MRI or follow-up.
* Use of investigational drugs within one month prior to enrollment or during the study.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults aged 55 to 90 years at the study center, including CN individuals, participants with MCI, and patients diagnosed with AD according to standardized criteria. All participants will undergo comprehensive cognitive assessment, neuroimaging, and biospecimen collection, and will be followed longitudinally for at least four years.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Regional Brain Sodium Concentration (mmol/L) Measured by 7 T ²³Na-MRI | Baseline to 1 year
  Quantitative regional brain sodium concentration measured by 7 T sodium (²³Na) MRI; units mmol/L; higher values indicate increased sodium concentration.
Change from Baseline in Resting-State Fractional Amplitude of Low-Frequency Fluctuations（fALFF, unitless) Measured by 7 T fMRI | baseline to 1year
  Fractional Amplitude of fALFF averaged within gray-matter mask (unitless; higher = greater spontaneous activity).
Change from Baseline in Mean Apparent Diffusion Coefficient (ADC) (×10-³ mm²/s) Derived from Dynamic Diffusion-Weighted Imaging (DynDWI) | Baseline to 1 year
  Mean ADC (×10-³ mm²/s) derived from DynDWI; higher values indicate increased diffusivity.
Change From Baseline in Fractional Anisotropy (FA, unitless) | Baseline to 1 year
  Change from baseline in DTI-derived FA values in major white matter tracts; higher FA indicates greater microstructural integrity.
Change From Baseline in Mean Diffusivity (MD, ×10-³ mm²/s) | Baseline to 1 year
  Change from baseline in DTI-derived MD values in major white-matter tracts; higher MD indicates increased water diffusivity (×10-³ mm²/s).

SECONDARY OUTCOMES:
Change from Baseline in Montreal Cognitive Assessment (MoCA) Total Score (0-30, points) | Baseline to 1 year
  Higher scores indicate better global cognition.
Change from Baseline in Clinical Dementia Rating (CDR) Global Score (0-3, points) | Baseline to 1 year
  Higher scores indicate more severe dementia.
Change from Baseline in Mini-Mental State Examination (MMSE) Total Score (0-30, points) | Baseline to 1 year
  Lower scores indicate greater impairment.
Change From Baseline of the Auditory Verbal Learning Test (AVLT) Total Learning Score | baseline to 1year
  AVLT total learning score is the sum of Trials N1-N6 (each trial scored 0-15; total range 0-90); higher scores indicate better verbal memory.
Change from Baseline in Rey-Osterrieth Complex Figure Test (ROCF) Combined Recall Score (0-72, points) | baseline to 1year
  Combined Recall = Immediate Recall (0-36) + Delayed Recall (0-36), scored with the 36-point Osterrieth method; range 0-72. Higher scores indicate better visuospatial (visual) memory.
Change From Baseline of the Clock Drawing Test (CDT) Score (0-5, points) | Baseline to 1 year
  CDT score ranges 0-5; higher scores indicate better visuospatial and executive function.
Change From Baseline of the Boston Naming Test (BNT) Total Score (0-60, points) | Baseline to 1 year
  BNT total score ranges 0-60; higher scores indicate better confrontational naming ability.
Change from Baseline in Digit Span Test (DST) Total Score (0-15, points) | Baseline to 1 year
  Forward (0-8) + backward (0-7); higher = better attention/working memory.
Change from Baseline in Symbol Digit Modalities Test (SDMT) Total Score (correct matches per 90 s) | Baseline to 1 year
  SDMT total score is the number of correct symbol-digit matches in 90 seconds (typical range 0-110); higher scores indicate better processing speed and attention.
Change from Baseline in Stroop Color-Word Test (SCWT) Incongruent Condition Completion Time (seconds) | Baseline to 1 year
  Shorter time indicates better cognitive flexibility and inhibition.
Change from Baseline in Neuropsychiatric Inventory (NPI) Total Score (0-144, points) | Baseline to 1 year
  NPI total score ranges 0-144; higher scores indicate more severe neuropsychiatric symptoms.
Change from Baseline in Hamilton Anxiety Rating Scale (HAMA) Total Score (0-56, points) | Baseline to 1 year
  HAMA total score ranges 0-56; higher scores indicate more severe anxiety symptoms.
Change from Baseline in Hamilton Depression Rating Scale (HAMD) Total Score (0-52, points) | Baseline to 1 year
  HAMD total score ranges 0-52; higher scores indicate more severe depressive symptoms.
Change from Baseline in Symptom Checklist-90 (SCL-90) Total Score (90-450, points) | Baseline to 1 year
  SCL-90 total score ranges 90-450; higher scores indicate greater overall psychological distress.
Change from Baseline in Activities of Daily Living (ADL) Scale Score (0-100, points) | Baseline to 1 year
  ADL total score ranges 0-100; higher scores indicate greater independence in basic self-care tasks.
Change from Baseline in Pittsburgh Sleep Quality Index (PSQI) Total Score (0-21, points) | Baseline to 1 year
  PSQI total score ranges 0-21; higher scores indicate poorer sleep quality over the past month
Change from Baseline in Trail Making Test (TMT) B-A Difference Score (seconds) | Baseline to 1 year
  Difference score calculated as Part B completion time minus Part A completion time (in seconds). Lower scores indicate better executive function after adjusting for processing speed.
Plasma Biomarkers of AD | Baseline to 1 year
  Percent changes from baseline in: amyloid-beta 40 and 42 (Aβ40, Aβ42), phosphorylated tau 181 and 217 (p-tau181, p-tau217) and neurofilament light (NfL); concentrations in pg/mL.
Change from Baseline in Hippocampal Volume (mm³) by FreeSurfer | Baseline to 1 year
  Bilateral hippocampal volume segmented with FreeSurfer; units mm³.
Number of participants with new cerebral microbleeds detected by susceptibility-weighted imaging (SWI) | Baseline to 1 year
  New microbleeds are defined as the appearance of ≥1 new hypointense lesion on SWI compared to baseline.
Change from Baseline in Brain Perivascular Spaces (PVS) Burden (semi-quantitative score) | Baseline to 1 year
  Description: PVS scored 0-4 in basal ganglia and 0-4 in centrum semiovale on 7 T MRI; global burden is the sum (0-8); higher scores indicate greater PVS load.

OTHER OUTCOMES:
apolipoprotein E (APOE) genotype (ε4 carrier status) | Baseline
  Proportion of participants carrying at least one ε4 allele of the APOE gene.
Identification of genetic susceptibility loci by genome-wide association study (GWAS) | Baseline
  Number and genomic location of susceptibility loci associated with Alzheimer's disease, as identified by GWAS.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided